CLINICAL TRIAL: NCT02107833
Title: A Phase 1, Randomized, Parallel-Design, Open-Label Study to Evaluate the Safety and Pharmacokinetics of Oral OPRX-106 (TNFR-Fc Fusion Protein) in Healthy Volunteers
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of Oral OPRX-106 (TNFR-Fc Fusion Protein) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protalix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB-106-001
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Human Volunteer
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 mg (Experimental): OPRX-106 2 mg oral once daily for 5 days
  Interventions: Drug: OPRX-106
- 8 mg (Experimental): OPRX-106 8 mg oral once daily for 5 days
  Interventions: Drug: OPRX-106
- 16 mg (Experimental): OPRX-106 16 mg oral once daily for 5 days
  Interventions: Drug: OPRX-106

INTERVENTIONS:
Drug: OPRX-106
  Other Names: TNF receptor-Fc fusion protein (TNFR-Fc)

SUMMARY:
: This is a Phase I, study to evaluate the safety and pharmacokinetics of oral OPRX-106 in healthy volunteers. Up to 18 healthy male subjects (age 18 years and older) will be randomized to one of three dose cohorts (up to 6 subjects per cohort), receiving OPRX-106 doses equivalent to 2mg, 8mg or 16mg Tumor Necrosis Factor receptor-Fc fusion protein. Subjects will receive once daily oral administrations of OPRX-106 for 5 consecutive days. Subjects will remain at the clinical center for 24 hours after the first administration (Day 1) of OPRX-106 including PK sampling and then return to the site daily for additional administrations and study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male age 18-45
* Body mass index (BMI) 18-30 kg/m2
* Male subjects or their partners must use an adequate method of contraception at all times during the study.
* Negative laboratory tests for HIV, HBcAb and HCV at the screening visit
* Naïve to any previous recombinant protein therapy
* Provide written informed consent
* Have the ability to understand the requirements of the study and to comply with the study protocol and dosing regimen

Exclusion Criteria:

* Clinical evidence of any active significant disease that could potentially compromise the ability of the Investigator to evaluate or interpret the effects of the study treatment on safety assessment, thus increasing the risk to the subject to unacceptable levels
* Presence of any acute or chronic diseases
* History of any allergies or protein-drug hypersensitivity
* Exposure to long-term steroid treatment within the last 12 months prior to the study
* Subject had a major operation in last 6 months
* Subject has received immunosuppressive treatment prior to the study
* Chronic use of any medication including vitamins
* Participation in another clinical trial during the previous 3 months (subject report)
* Reported history of alcohol or drug abuse
* Subjects with short bowel (more than 1 m removed of small bowel).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 5 days
  Adverse events from subject reporting or other assessments

SECONDARY OUTCOMES:
Area under the curve | 24 hours
  OPRX-106 concentrations measured at 0, 2, 4, 6, 8,10, 12, 14, 16 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Einat Almon, PdH, Study Director — Protalix Ltd.
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel